CLINICAL TRIAL: NCT05286905
Title: Biomechanical Testing, Finite Element Analysis and Pilot, Prospective, Randomized, Experimental Clinical Study of Osteosynthesis of Reverse Oblique Peritrochanteric Fractures With PFLP vs Cephalomedullary Nail.
Brief Title: FEA, Biomechanical and Clinical Study of R.O. Peritrochanteric Fractures With PFLP vs Cephalomedullary Nail.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University General Hospital of Patras (Other)
Responsible Party: Principal Investigator, Parchas Nikolaos, Md. Resident, Department of Orthopedics and Traumatiology, University General Hospital of Patras, University General Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13474
Record Dates: First submitted 2022-02-27; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Pertrochanteric Fracture of Femur, Closed
Keywords: Peritrochanteric fractures; reverse oblique; proximal femur locking plate; Cephalomedullary nail

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who receive cephalomedullary nail (Active Comparator): Patients who receive cephalomedullary nail
  Interventions: Device: Osteosynthesis cephalomedullary nail
- Patients who receive proximal femur locking plate (Active Comparator): Patients who receive proximal femur locking plate
  Interventions: Device: Osteosynthesis proximal femur locking plate

INTERVENTIONS:
Device: Osteosynthesis cephalomedullary nail — Osteosynthesis of reverse oblique peritrochanteric fractures with cephalomedullary nail
  Arms: Patients who receive cephalomedullary nail
Device: Osteosynthesis proximal femur locking plate — Osteosynthesis of reverse oblique peritrochanteric fractures with proximal femur locking plate
  Arms: Patients who receive proximal femur locking plate

SUMMARY:
Hip fractures are the second most common fracture regardless of age, while at the same time its incidence is on the rise and it is expected to keep increasing in the future. In addition, hip fractures oppose a serious problem for both patients and clinicians, as they are associated with high rates of morbidity, reduced quality of life, impeded independent functionality and higher institutionalization rates. Several osteosynthesis techniques have been proposed for surgical correction of hip fractures which can be grouped into 3 main categories: a) Dynamic Hip Screw (DHS) extramedullary systems, b) Proximal femoral nail N [PN] PFNA], γ-nail [GN] or other implants) and (c) Dynamic Condylar Screw, Angled blade plates, Proximal Femur Locking Plate (PFLP).

This study will compare the use of anatomical proximal femur locking plates ( PeriLock, Smith& Nephew) with an intramedullary nailing system, one of the most common and literature supported implants for the reduction of reverse oblique intertrochanteric fractures, classified as A31- 1,3 according to AO. The study will include Biomechanical testing and finite element analysis of the implants in an experimental setup using artificial bones performed at the Laboratory of Technology and Strength of Materials of the Department of Mechanical Engineering and Aeronautics of the University of Patras. and a pilot, prospective, randomized clinical study in a sample of 30 patients divided into 2 groups, where comparison of perioperative and intraoperative data will be accessed.

The purpose of this study is to evaluate the efficacy and mechanical stability as wells as the clinical and radiological parameters as well as quality-of-life indicators in patients with reverse oblique hip fractures The primary goal of to investigate whether there are statistically significant differences in the main radiological parameters (cut-out, misalignment of the femoral head, loss of alignment, defective posture, non-union), while The second primary goal is to assess the functional and general health status of patients up to 24 weeks postoperatively, using special clinical evaluation scales (Harris Hip score-HHS and Oxford hip score-OHS), as well as pain levels perioperatively

DETAILED DESCRIPTION:
Background Hip fractures are the second most common fractures regardless of age . At the same time, the prevalence of these fractures is increasing, with the total number of admissions for hip fractures in the US is estimated to reach 289,000 by 2030 with an increase to 4.5 million by 2050. In the United Kingdom, although there has been an age-weighted decline in hip fractures of 0.5% per year, it is estimated that their incidence in the United Kingdom will double in the next 25 years. In addition, hip fractures are associated with a high risk of mortality, especially in the elderly, as well as reduced mobility. Their consequences in the elderly are significant due primarily to the increased mortality and secondarily to the negative effects on the health of patients resulting in reduced mobility and influence of their quality of life. In a recent review of 38 studies by Dyer et al, hip fracture survivors had significantly affected mobility, independent functionality, health, quality of life, and higher institutionalization rates compared to their respective age control group without fracture. Even with advances in rehabilitation institutes and new scientific protocols for the optimal treatment of hip fragility fractures, the in-hospital mortality rate was 2.4% and the overall mortality, one year postoperatively, was 18.7% and complete recovery or slight reduction of mobility was achieved in 32.1% of patients. In a recent study by the Swedish Hip Fracture Registry, the first-year mortality rate was about 20% for women and 30% for men in a total population study of 289,603 patients with first hip fracture. during a period of 20 years (1998-2017).

The first mobilization after a hip fracture seems to be beneficial for patients as it is associated with reduced complications due to prolonged bed rest and helps the fracture heal. Consequently, the vast majority of fractures require surgical interventions to allow for fast mobilization and loading of the limb. Various osteosynthesis techniques have been proposed and used which fall into three main categories: a) Dynamic Hip Screw (DHS) extramedullary systems, b) Proximal femoral nail N [PN] PFNA], γ-nail [GN] or other implants) and (c) Dynamic Condylar Screw, Angled blade plates, Proximal Femur Locking Plate (PFLP). The type of osteosynthesis is based on the pattern of the fracture, the characteristics of the patient and the preference of the surgeon In our study we will analyze the lateral oblique (reverse oblique) peritrochanteric fractures that are classified as A31-1,2,3 according to AO and extend on the lateral wall of the proximal femur (Figure 1).

In this fracture category we will compare the anatomical locked plate PERI-LOC◊ 4.5mm Proximal Femur Locking Plate (PFLP) (Smith & Nephew) with cephalomedullary nail [Figure 2]. PFLP is an implant characterized by the ability to place multiple screws in both the head (5) and the femoral diaphysis. It also has an anatomical design, offers immediate reduction of the fracture with the possibility of additional placement of wires while there is a special guide for the transdermal placement of the peripheral screws. In contrast, the cephalic nails, using a transverse screw compressor, allow the linear compression of the descending sections, while providing a high degree of rotational stability.

The common problem with cephalic nails is that they cannot usually align the outwardly displaced central part of the head (Figure 2) and in addition, the posterior slip of the transverse screw is parallel to the fracture line and exacerbates postoperative misalignment. during charging. Biomechanically, however, it is the central part of the nail that resists the sliding forces and holds the further displacement of the fracture. According to the existing literature, there are conflicting data on the stability of PFLP's. Ozkan et al. In a biomechanical study on the stability of PFLPs against intramedullary nails for unstable intertrochanteric fractures (but not reverse oblique ones) they concluded that for subtrochanteric fractures, PFLP's provided greater stability, but the difference was not statistically significant. A retrospective study of the efficacy of PFLP in peritchanteric fractures has shown that it has fewer complications than other methods. At the same time, biomechanical studies suggest that the axial stability of PFLP'S is less than that of intramedullary implants. In studies evaluating the postoperative parameters of peritrochanteric fractures, good results have been reported in terms of anatomical reduction, fracture healing and patient function scores. Nevertheless, it is shown that the intramedullary nails offer greater mechanical stiffness, stabilization and shorter time of onset of porous. It should be noted, however, that a direct comparison of the peri-loc plate with the cephalomedullary nails is not known to have been published in the literature regarding unstable subtrochanteric fractures, while in a study comparing them biomechanically it appears that this material has comparable stability with the TIT (Smith and Nephew) nail.

I. CLINICAL STUDY Purpose of the study The proposed pilot, monocentric, randomized controlled trial is designed to evaluate clinical and radiological parameters as well as quality-of-life indicators in patients with reverse oblique hip fractures (A31-1.3 against AO) undergoing surgery. With the anatomical proximal femur locking plate, against an intermedullary nailing system. Our main assumption is that the plate will provide better radiological and possibly better clinical results compared to the intramedullary nailing system. The biomechanical differences of the two implants will be examined in the biomechanical study.

Primary objective The primary goal of this study is to investigate whether there are statistically significant differences in the main radiological parameters (cut-out, misalignment of the femoral head, loss of alignment, defective posture, non-union), in patients over 65 years of age with reverse oblique hip fractures treated with the classic intramedullary nail system versus PFLP over a 24-week follow-up period.

The second primary goal is to assess the functional status of patients up to 24 weeks postoperatively, using special clinical evaluation scales (Harris Hip score-HHS and Oxford hip score-OHS).

Sub-objectives

Several sub-objectives will also be studied in order to evaluate the efficacy and safety of the above implants, quantifying and drawing evidence from the observed differences between the control groups in the following:

1. Comparison of perioperative and intraoperative surgical data (surgery delay, age-adjusted Carlson comorbidity index, operating time, radioscopy time and dosage, blood loss, length of hospital stay, total dose of analgesics per class of drug (Dual Energy X-ray Absorptiometry) of the healthy hip, the time of fracture healing, the intraoperative complications that depend on the surgeon's manipulations, such as incorrect placement of the compression screw, fracture extension, non-anatomical reduction, osteosynthesis in varus/valgus position, or rotational deformity as well as the assessment of radiological parameters such as the TAD index using postoperative pelvic computed tomography).
2. Quantitative assessment of pain during the perioperative period and at 6, 12 and 24 weeks postoperatively, using the visual analogue scale.
3. Assessment of the patient's general health status before surgery and at 6, 12 and 24 weeks postoperatively using the SF-36 assessment form, the EQ-5D-3L questionnaire, the SARC-F index and the elderly mobility scale (EMS).

Patient selection criteria.

1. A31-1,3 intertrochanteric fracture (AO classification) due to trauma, closed injury
2. Patients over 65 years of age
3. Presentation in the hospital within 7 days from the
4. There are no concomitant injuries or previous operations on the unaffected hip

Patient exclusion criteria

1. Patients with concomitant injuries that affect the treatment and rehabilitation of the affected limb
2. Patients with associated neurovascular injuries requiring immediate surgery
3. Patients with limited Greek language proficiency, including family members
4. Patients who refuse to sign admission consent to the study
5. Patients with severe dementia, bedridden and severe comorbidities that are a contraindication to surgery

Sample size - Statistical analysis This study will use two primary efficacy scales, the Oxford Hip Score and the Harris Hip Score. Minimum clinically significant differences for HHS have been estimated between 7 and 10, while for OHS between 5 and 7. The aim will be to evaluate 15 patients in each group, as this will provide a sufficient sample for 90% strength and for two primary outcome measures. With a projected abandonment rate of 15%, the total number of patients required will be 35. If collection proves problematic during the study, then the target will be reduced and the more common 80% power level will be considered sufficient. For this scenario, the total number of patients required will be 35 (including the 15% non-completion of the study).

The main outcome measure of radiological failure is a binary result (failure / failure). A binary regression accounting model will be performed to estimate the correlation between the 'failure' outcome and the implant type (PFLP, TIT). The complication rate of PFLP versus nail at 24 weeks postoperatively will be compared using the x2 test (with a significance level of 5%). Differences between HHS and OHS between groups will be assessed using the t-test for independent variables at 24 weeks postoperatively with a significance level of 5%. Test levels will be adjusted using Holm-Bonferroni methods to allow multiple comparisons. A linear regression analysis will also be used to quantify the effects of treatment methods on each of the primary outcome measures, after weighing the effects of other important, potentially confusing factors (eg age, gender) recorded for each patient.

II. BIOMECHANICAL STUDY AND ANALYSIS OF PASSED DATA

The experimental test will be performed at the Laboratory of Technology and Strength of Materials of the Department of Mechanical Engineering and Aeronautics of the University of Patras. Two systems of intramedullary implants will be used, the anatomically locked plate PERI-LOC 4.5mm Proximal Femur Locking Plate (S & N) and a cephalomedullary nailing system.

Our hypothesis is based on the fact that the individual differences between the two osteosynthesis systems for the treatment of two-way fractures may create different patterns of deformation distribution and, consequently, dissimilar biomechanical behaviors. For the purpose of the study, synthetic osteoporotic femurs will be used in which, through osteotomies, the experimental model of an unstable fracture will be created. This will be followed by osteosynthesis of the fracture with the osteostabilization systems under study. The correctness of the implantation of the studied intramedullary systems in the synthetic femurs will be checked radiologically. The implanted bones will be placed in a suitable device, where a static charge will be applied. The induced deformity will be evaluated as it is distributed over the entire surface of the proximal femur with the method of digital image correlation (Digital Image Correlation-DIC) but also the maximum load causing induction of osteosynthesis failure.

In addition to the experimental studies, the biomechanical behavior of the implants under study will be studied using the finite element method. To this end, parametric finite element models of the descending femur and intramedullary implants will be developed. These models, once validated by the mechanical tests, will be used to evaluate possible biomechanical system failure scenarios by performing a detailed bone and/or implant failure analysis.

ELIGIBILITY:
Inclusion Criteria:

1. A31-1,3 intertrochanteric fracture ( AO classification) due to trauma, closed injury.
2. Patients over 65 years of age
3. Presentation in the hospital within 7 days from the fracture
4. There are no concomitant injuries or previous operations on the unaffected hip

Exclusion Criteria:

1. Patients with concomitant injuries that affect the treatment and rehabilitation of the affected limb
2. Patients with associated neurovascular injuries requiring immediate surgery
3. Patients with limited Greek language proficiency, including family members
4. Patients who refuse to sign admission consent to the study
5. Patients with severe dementia, bedridden and severe comorbidities that are a contraindication to surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-10-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Radiological differences of cephalodullary nail vs PFLP | 24-week follow-up period
  tatistically significant differences in the main radiological parameters (cut-out, misalignment of the femoral head, loss of alignment, defective posture, non-union), in patients over 65 years of age with reverse oblique hip fractures treated with the classic intramedullary nail system versus PFLP over a .
Functional status (Oxford hip score-OHS) | 24 weeks
  Assess the functional status of patients up to 24 weeks postoperatively

SECONDARY OUTCOMES:
Functional status (Harris Hip score-HHS) | 24 weeks
  Assess the functional status of patients up to 24 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Panagopoulos, As. Prof., Study Director — University of Patras
Locations (1):
- General University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Yes
Patients personal information will NOT be shared, radiographic, statistical and score data will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the completion of the study
Access Criteria: Free

REFERENCES:
- [Background] Bergh C, Wennergren D, Moller M, Brisby H. Fracture incidence in adults in relation to age and gender: A study of 27,169 fractures in the Swedish Fracture Register in a well-defined catchment area. PLoS One. 2020 Dec 21;15(12):e0244291. doi: 10.1371/journal.pone.0244291. eCollection 2020. PMID 33347485
- [Background] Stevens JA, Rudd RA. The impact of decreasing U.S. hip fracture rates on future hip fracture estimates. Osteoporos Int. 2013 Oct;24(10):2725-8. doi: 10.1007/s00198-013-2375-9. Epub 2013 Apr 30. PMID 23632827
- [Background] White SM, Griffiths R. Projected incidence of proximal femoral fracture in England: a report from the NHS Hip Fracture Anaesthesia Network (HIPFAN). Injury. 2011 Nov;42(11):1230-3. doi: 10.1016/j.injury.2010.11.010. Epub 2010 Dec 22. PMID 21183180
- [Background] Veronese N, Maggi S. Epidemiology and social costs of hip fracture. Injury. 2018 Aug;49(8):1458-1460. doi: 10.1016/j.injury.2018.04.015. Epub 2018 Apr 20. PMID 29699731
- [Background] Dyer SM, Crotty M, Fairhall N, Magaziner J, Beaupre LA, Cameron ID, Sherrington C; Fragility Fracture Network (FFN) Rehabilitation Research Special Interest Group. A critical review of the long-term disability outcomes following hip fracture. BMC Geriatr. 2016 Sep 2;16(1):158. doi: 10.1186/s12877-016-0332-0. PMID 27590604
- [Background] Wang J, Ma JX, Jia HB, Chen Y, Yang Y, Ma XL. Biomechanical Evaluation of Four Methods for Internal Fixation of Comminuted Subtrochanteric Fractures. Medicine (Baltimore). 2016 May;95(19):e3382. doi: 10.1097/MD.0000000000003382. PMID 27175636
- [Background] Karagiannis A, Papakitsou E, Dretakis K, Galanos A, Megas P, Lambiris E, Lyritis GP. Mortality rates of patients with a hip fracture in a southwestern district of Greece: ten-year follow-up with reference to the type of fracture. Calcif Tissue Int. 2006 Feb;78(2):72-7. doi: 10.1007/s00223-005-0169-6. Epub 2006 Feb 6. PMID 16467975
- [Background] Civinini R, Paoli T, Cianferotti L, Cartei A, Boccaccini A, Peris A, Brandi ML, Rostagno C, Innocenti M. Functional outcomes and mortality in geriatric and fragility hip fractures-results of an integrated, multidisciplinary model experienced by the "Florence hip fracture unit". Int Orthop. 2019 Jan;43(1):187-192. doi: 10.1007/s00264-018-4132-3. Epub 2018 Aug 29. PMID 30159804
- [Background] Meyer AC, Ek S, Drefahl S, Ahlbom A, Hedstrom M, Modig K. Trends in Hip Fracture Incidence, Recurrence, and Survival by Education and Comorbidity: A Swedish Register-based Study. Epidemiology. 2021 May 1;32(3):425-433. doi: 10.1097/EDE.0000000000001321. PMID 33512961
- [Background] Papasimos S, Koutsojannis CM, Panagopoulos A, Megas P, Lambiris E. A randomised comparison of AMBI, TGN and PFN for treatment of unstable trochanteric fractures. Arch Orthop Trauma Surg. 2005 Sep;125(7):462-8. doi: 10.1007/s00402-005-0021-5. PMID 16059696
- [Background] Kim JW, Oh CW, Byun YS, Oh JK, Kim HJ, Min WK, Park SK, Park BC. A biomechanical analysis of locking plate fixation with minimally invasive plate osteosynthesis in a subtrochanteric fracture model. J Trauma. 2011 Jan;70(1):E19-23. doi: 10.1097/TA.0b013e3181d40418. PMID 20495493
- [Background] Socci AR, Casemyr NE, Leslie MP, Baumgaertner MR. Implant options for the treatment of intertrochanteric fractures of the hip: rationale, evidence, and recommendations. Bone Joint J. 2017 Jan;99-B(1):128-133. doi: 10.1302/0301-620X.99B1.BJJ-2016-0134.R1. PMID 28053268
- [Background] Knobe M, Gradl G, Buecking B, Gackstatter S, Sonmez TT, Ghassemi A, Stromps JP, Prescher A, Pape HC. Locked minimally invasive plating versus fourth generation nailing in the treatment of AO/OTA 31A2.2 fractures: A biomechanical comparison of PCCP((R)) and Intertan nail((R)). Injury. 2015 Aug;46(8):1475-82. doi: 10.1016/j.injury.2015.05.011. Epub 2015 May 14. PMID 25997559
- [Background] Serrano R, Blair JA, Watson DT, Infante AF Jr, Shah AR, Mir HR, Maxson BJ, Downes KL, Sanders RW. Cephalomedullary Nail Fixation of Intertrochanteric Femur Fractures: Are Two Proximal Screws Better Than One? J Orthop Trauma. 2017 Nov;31(11):577-582. doi: 10.1097/BOT.0000000000000967. PMID 28827501
- [Background] Ozkan K, Turkmen I, Sahin A, Yildiz Y, Erturk S, Soylemez MS. A biomechanical comparison of proximal femoral nails and locking proximal anatomic femoral plates in femoral fracture fixation: A study on synthetic bones. Indian J Orthop. 2015 May-Jun;49(3):347-51. doi: 10.4103/0019-5413.156220. PMID 26015637
- [Background] Polat G, Akgul T, Ekinci M, Bayram S. A biomechanical comparison of three fixation techniques in osteoporotic reverse oblique intertrochanteric femur fracture with fragmented lateral cortex. Eur J Trauma Emerg Surg. 2019 Jun;45(3):499-505. doi: 10.1007/s00068-018-1061-1. Epub 2019 Jan 2. PMID 30600335
- [Background] Ibrahim S, Meleppuram JJ. A retrospective analysis of surgically-treated complex proximal femur fractures with proximal femoral locking compression plate. Rev Bras Ortop. 2017 Jan 7;52(6):644-650. doi: 10.1016/j.rboe.2016.12.012. eCollection 2017 Nov-Dec. PMID 29234646
- [Background] Collinge CA, Hymes R, Archdeacon M, Streubel P, Obremskey W, Weber T, Watson JT, Lowenberg D; Members of the Proximal Femur Working Group of the Southeast Trauma Consortium. Unstable Proximal Femur Fractures Treated With Proximal Femoral Locking Plates: A Retrospective, Multicenter Study of 111 Cases. J Orthop Trauma. 2016 Sep;30(9):489-95. doi: 10.1097/BOT.0000000000000602. PMID 27144821
- [Background] Walmsley D, Nicayenzi B, Kuzyk PR, Machin A, Bougherara H, Schemitsch EH, Zdero R. Biomechanical analysis of the cephalomedullary nail versus the trochanteric stabilizing plate for unstable intertrochanteric femur fractures. Proc Inst Mech Eng H. 2016 Dec 1;230(12):1133-1140. doi: 10.1177/0954411916676508. Epub 2016 Oct 26. PMID 27789875
- [Background] Viberg B, Rasmussen KMV, Overgaard S, Rogmark C. Poor relation between biomechanical and clinical studies for the proximal femoral locking compression plate. Acta Orthop. 2017 Aug;88(4):427-433. doi: 10.1080/17453674.2017.1304207. Epub 2017 Mar 13. PMID 28287002
- [Background] Singh AK, Narsaria N, Gupta RK. A biomechanical study comparing proximal femur nail and proximal femur locking compression plate in fixation of reverse oblique proximal femur fractures. Injury. 2017 Oct;48(10):2050-2053. doi: 10.1016/j.injury.2017.05.029. Epub 2017 May 22. PMID 28801202
- [Background] Kumar N, Kataria H, Yadav C, Gadagoli BS, Raj R. Evaluation of proximal femoral locking plate in unstable extracapsular proximal femoral fractures: Surgical technique & mid term follow up results. J Clin Orthop Trauma. 2014 Sep;5(3):137-45. doi: 10.1016/j.jcot.2014.07.009. Epub 2014 Sep 10. PMID 25983487
- [Background] Shah MD, Kapoor CS, Soni RJ, Patwa JJ, Golwala PP. Evaluation of outcome of proximal femur locking compression plate (PFLCP) in unstable proximal femur fractures. J Clin Orthop Trauma. 2017 Oct-Dec;8(4):308-312. doi: 10.1016/j.jcot.2016.11.005. Epub 2016 Nov 21. PMID 29062210
- [Background] Hu SJ, Zhang SM, Yu GR. Treatment of femoral subtrochanteric fractures with proximal lateral femur locking plates. Acta Ortop Bras. 2012 Dec;20(6):329-33. doi: 10.1590/S1413-78522012000600003. PMID 24453626
- [Background] Zha GC, Chen ZL, Qi XB, Sun JY. Treatment of pertrochanteric fractures with a proximal femur locking compression plate. Injury. 2011 Nov;42(11):1294-9. doi: 10.1016/j.injury.2011.01.030. Epub 2011 Feb 26. PMID 21356535
- [Background] Zubairi A, Rashid RH, Zahid M, Hashmi PM, Noordin S. Proximal Femur Locking Plate for Sub-Trochanteric Femur Fractures: Factors Associated with Failure. Open Orthop J. 2017 Aug 29;11:1058-1065. doi: 10.2174/1874325001711011058. eCollection 2017. PMID 28979608
- [Background] Arirachakaran A, Amphansap T, Thanindratarn P, Piyapittayanun P, Srisawat P, Kongtharvonskul J. Comparative outcome of PFNA, Gamma nails, PCCP, Medoff plate, LISS and dynamic hip screws for fixation in elderly trochanteric fractures: a systematic review and network meta-analysis of randomized controlled trials. Eur J Orthop Surg Traumatol. 2017 Oct;27(7):937-952. doi: 10.1007/s00590-017-1964-2. Epub 2017 Apr 22. PMID 28434124
- [Background] Dhamangaonkar AC, Joshi D, Goregaonkar AB, Tawari AA. Proximal femoral locking plate versus dynamic hip screw for unstable intertrochanteric femoral fractures. J Orthop Surg (Hong Kong). 2013 Dec;21(3):317-22. doi: 10.1177/230949901302100311. PMID 24366792
- [Background] Lee WT, Murphy D, Kagda FH, Thambiah J. Proximal femoral locking compression plate for proximal femoral fractures. J Orthop Surg (Hong Kong). 2014 Dec;22(3):287-93. doi: 10.1177/230949901402200304. PMID 25550004
- [Background] Agrawal P, Gaba S, Das S, Singh R, Kumar A, Yadav G. Dynamic hip screw versus proximal femur locking compression plate in intertrochanteric femur fractures (AO 31A1 and 31A2): A prospective randomized study. J Nat Sci Biol Med. 2017 Jan-Jun;8(1):87-93. doi: 10.4103/0976-9668.198352. PMID 28250681
- [Background] Streubel PN, Moustoukas M, Obremskey WT. Locked plating versus cephalomedullary nailing of unstable intertrochanteric femur fractures. Eur J Orthop Surg Traumatol. 2016 May;26(4):385-90. doi: 10.1007/s00590-016-1743-5. Epub 2016 Feb 26. PMID 26920361
- [Background] He S, Yan B, Zhu J, Huang X, Zhao J. High failure rate of proximal femoral locking plates in fixation of trochanteric fractures. J Orthop Surg Res. 2018 Oct 5;13(1):248. doi: 10.1186/s13018-018-0951-6. PMID 30290848
- [Background] Han L, Liu JJ, Hu YG, Quan RF, Fang WL, Jin B, Lin WL. Controlled study on Gamma nail and proximal femoral locking plate for unstable intertrochanteric femoral fractures with broken lateral wall. Sci Rep. 2018 Jul 24;8(1):11114. doi: 10.1038/s41598-018-28898-6. PMID 30042398
- [Background] Hodel S, Beeres FJP, Babst R, Link BC. Complications following proximal femoral locking compression plating in unstable proximal femur fractures: medium-term follow-up. Eur J Orthop Surg Traumatol. 2017 Dec;27(8):1117-1124. doi: 10.1007/s00590-017-1981-1. Epub 2017 May 25. PMID 28547675